CLINICAL TRIAL: NCT00480636
Title: Fragmin Safety And Efficacy In The Treatment Of Acute Deep-Vein Thrombosis With Or Without Pulmonary Embolism And Extended Thromboprophylaxis In Cancer Patients In Slovakia (An Open, Prospective, Non-Comparative Study)
Brief Title: Fragmin In The Treatment Of Acute Deep-Vein Thrombosis With Or Without Pulmonary Embolism In Cancer Patients
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Other Study IDs: A6301082
Record Dates: First submitted 2007-05-29; First posted 2007-05-31 (Estimated); Results first posted 2010-08-10 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-07

CONDITIONS: Acute Deep Vein Thrombosis
MeSH Terms: interventions — Dalteparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- One cohort of patients treated with dalteparin.: About 100 patients with deep-vein thrombosis and with or without pulmonary embolism will be included in the study.
  Interventions: Drug: Fragmin (dalteparin sodium )

INTERVENTIONS:
Drug: Fragmin (dalteparin sodium ) — Month 1: dalteparin 200 IU/kg SC once daily. Months 2-6: dalteparin 150 IU/kg SC, once daily.
  Other Names: Fragmin

SUMMARY:
To collect postmarketing data about Fragmin safety and efficacy in the treatment of deep vein thrombosis with or without pulmonary embolism in cancer patients.

DETAILED DESCRIPTION:
Method: consecutive patient sampling. Patients were (are) included in the study in consecutive manner if they fulfilled the inclusion criteria and any of the exclusion criteria were not present.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient of 18 - 70 years of age.
* Cancer patient with proven deep-vein thrombosis with or without pulmonary embolism confirmed by combination of clinical signs and symptoms, pulmonary hypertension on echocardiogram, X-ray examination of the lung and eventually perfusion/ventilation scan of the lung.

Exclusion Criteria:

* Bleeding
* Hypersensitivity to FRAGMIN® or other low-molecular weight heparins.
* Serum creatinine level > 150 umol/l.
* Platelet count of less than 100 000 per cubic millimeter at the beginning of the therapy.
* Patient on oral anticoagulation therapy in the last 7 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients are identified in primary care setting.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2007-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6301082&StudyName=Fragmin%20In%20The%20Treatment%20Of%20Acute%20Deep-Vein%20Thrombosis%20With%20Or%20Without%20Pulmonary%20Embolism%20In%20Cancer%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- Dalteparin: Dalteparin 200 International Units per kilogram (IU/kg) total body weight subcutaneously (SC) once daily (QD) for Month 1, then 150 IU/kg total body weight SC QD from Months 2 to 6.
Period: Overall Study
Arm/Group | Dalteparin
Started | 102
Completed | 83
Not Completed | 19
Not completed — Death | 12
Not completed — Lost to Follow-up | 4
Not completed — Other | 2
Not completed — Lost to follow-up; subsequently died | 1

BASELINE CHARACTERISTICS:
Groups:
- Dalteparin: Dalteparin 200 IU/kg total body weight SC QD for Month 1, then 150 IU/kg total body weight SC QD from Months 2 to 6.
Arm/Group | Dalteparin
Number analyzed (Participants) | 102
Age, Customized [Number; unit: Participants]
  Between 18 and 44 years | 4
  Between 45 and 64 years | 58
  >= 65 years | 39
  Unspecified | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 61.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Resolution of Deep Vein Thrombosis (DVT) of the Leg
Description: Resolution criteria: clinical cure, defined as negative results of a compressive ultrasound examination of the leg
Time Frame: Month 6 or End of Treatment (EOT) (up to Month 6)
Population: Full analysis set (FAS): all participants who received at least 1 dose of the study treatment and who had at least 1 post baseline efficacy measurement.
Measure: Number; unit: Participants
Arm/Group | Dalteparin
Number analyzed (Participants) | 102
Participants | 43

2. Secondary Outcome: Number of Participants With Severe Bleeding That Resulted in a Transfusion of at Least 2 Units of Blood
Description: Episodes of the severe bleeding (intracranial, intraspinal, intraocular, retroperitoneal, or in pericardial area) or bleeding from gastrointestinal (GIT), urinary system or gynecological bleeding resulted in a need for a transfusion of at least 2 units of blood. Subjects were assessed for severe bleeding as part of a systematic adverse event assessment.
Time Frame: Baseline through Month 6 or EOT (up to Month 6)
Population: The safety analysis set was defined as all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Dalteparin
Number analyzed (Participants) | 102
Participants | 0

3. Secondary Outcome: Number of Participants With Severe Bleeding That Resulted in a Decrease in Hemoglobin Level of at Least 2.0 Grams Per Deciliter (g/dL)
Description: Episodes of the severe bleeding (intracranial, intraspinal, intraocular, retroperitoneal, or in pericardial area) or bleeding from GIT, urinary system or gynecological bleeding which led to a drop of hemoglobin of at least 2.0 g/dL. Subjects were assessed for severe bleeding as part of a systematic adverse event assessment.
Time Frame: Baseline through Month 6 or EOT (up to Month 6)
Population: Safety analysis set.
Measure: Number; unit: Participants
Arm/Group | Dalteparin
Number analyzed (Participants) | 102
Participants | 0

4. Secondary Outcome: Percent of Participants With and Without Pulmonary Embolism (PE)
Description: PE (diagnosed on the basis of ventilation-perfusion scan of the lungs or autopsy)
Time Frame: Baseline, Week 2, Month 1, Month 3, and Month 6 or EOT (up to Month 6)
Population: FAS. n = number of participants per PE status at observation.
Measure: Number; unit: Percent of participants
Arm/Group | Dalteparin
Number analyzed (Participants) | 102
Percent of participants
  Baseline with PE (n = 16) | 15.7
  Baseline without PE (n = 82) | 80.4
  Baseline with missing information (n = 4) | 3.9
  Week 2 with PE (n = 7) | 6.9
  Week 2 without PE (n = 85) | 83.3
  Week 2 with missing information (n = 10) | 9.8
  Month 1 with PE (n = 3) | 2.9
  Month 1 without PE (n = 96) | 94.1
  Month 1 with missing information (n = 3) | 2.9
  Month 3 with PE (n = 1) | 1.0
  Month 3 without PE (n = 91) | 89.2
  Month 3 with missing information (n = 10) | 9.8
  Month 6 or EOT with PE (n = 3) | 2.9
  Month 6 or EOT without PE (n = 85) | 83.3
  Month 6 or EOT with missing information (n = 14) | 13.7

5. Secondary Outcome: Number of Participants With Recurrent DVT
Description: Defined as the number of participants with recurrence of DVT (diagnosed using compressive ultrasound examination or autopsy) after it has resolved (at the same location) or occurrence of new DVT at a new location on any of the post-baseline visits
Time Frame: Month 6 or EOT (up to Month 6)
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Dalteparin
Number analyzed (Participants) | 102
Participants | 3

ADVERSE EVENTS:
Arm/Group | Dalteparin
Serious Adverse Events (participants affected / at risk) | 13/102
Other Adverse Events (participants affected / at risk) | 0/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalteparin (N=102)
Cardiopulmonary failure (Cardiac disorders) | 2
Disease progression (General disorders) | 9
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Embolism (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.